CLINICAL TRIAL: NCT02813304
Title: Rest or Gradual Reloading in Acute Presentations of Rotator Cuff Tendinopathy - A Randomised Control Trial
Brief Title: Comparison of Two Treatments for Acute Rotator Cuff Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean-Sébastien Roy, Associate Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016- 494
Record Dates: First submitted 2016-06-21; First posted 2016-06-24 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2016-02

CONDITIONS: Acute Rotator Cuff Tendinopathy
Keywords: Acute; rotator cuff tendinopathy; exercise; loading; ice; cryotherapy; randomised control trial
MeSH Terms: conditions — Motor Activity | interventions — RE1-silencing transcription factor; Cryotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gradual reloading (Experimental): Participants will be asked to perform isometric strengthening exercises in lateral rotation and abduction (see Table 1). In a sitting position (with folded towel between body and arm), participants will place their affected arm by the side with the elbow gently tucked in close to the body, elbow flexed at 90°, and the thumb pointing upwards. The opposite hand (the uninvolved side) will resist the lateral rotation and abduction. They will be asked to push against the uninvolved hand, building up to sub-maximal pressure (approximately 50% to 75% of the maximum possible force; practice during the meeting with the treating physiotherapist using EMG recording) over five seconds.
  Interventions: Behavioral: Gradual reloading
- Rest and cryotherapy (Active Comparator): Participants will be asked to apply ice wrap on their painful shoulder 3 times a day over the area of pain for 15 minutes. They will be asked to place the ice wrap inside a damp towel cloth (minimise the risk of an ice burn) and secure around the shoulder with a towel. After the 15 minutes, they will be asked to perform gentle, slow, pain free shoulder movements that do not provoke pain. All participants will be provided with a commercial ice wrap and a towel cloth. They will also be asked to avoid painful movements, working above shoulder level, repeated or sustained elevation movements and lifting weights.
  Interventions: Behavioral: Rest and cryotherapy

INTERVENTIONS:
Behavioral: Gradual reloading — Participants will be asked to perform isometric strengthening exercises in lateral rotation and abduction. Participants will place their affected arm by the side with the elbow gently tucked in close to the body, elbow flexed at 90°, and the thumb pointing upwards. The opposite hand will resist the lateral rotation and abduction. They will be asked to push against the uninvolved hand, building up to sub-maximal pressure (approximately 50% to 75% of the maximum possible force) over five seconds. Then the contraction will be slowly released. A maximum pain level of 5/10 will be accepted when performing the contraction. Elevation movements will also be performed 3 times a day in the frontal, sagittal and scapular plane.
  Arms: Gradual reloading
Behavioral: Rest and cryotherapy — Participants will be asked to apply ice wrap on their painful shoulder 3 times a day over the area of pain for 15 minutes. They will be asked to place the ice wrap inside a damp towel cloth (minimise the risk of an ice burn) and secure around the shoulder with a towel. After the 15 minutes, they will be asked to perform gentle, slow, pain free shoulder movements that do not provoke pain. All participants will be provided with a commercial ice wrap. They will also be asked to avoid painful movements, working above shoulder level, repeated or sustained elevation movements and lifting weights.
  Arms: Rest and cryotherapy

SUMMARY:
The primary objective of this study is to compare the short-term effectiveness (2 and 6 weeks following the start of the rehabilitation program), in terms of symptoms and functional limitations, of a rehabilitation program centered on gradual reloading to a rehabilitation program centered on rest and cryotherapy in individuals with acute rotator cuff tendinopathy. The secondary objective is to explore the effects of these programs on shoulder control (acromiohumeral distance), subacromial structures (supraspinatus tendon thickness) and central pain modulation. The hypothesis is that the rehabilitation program centered on gradual reloading will lead to a faster improvement at week 2 and 6 when compared to the program centered on rest and cryotherapy.

DETAILED DESCRIPTION:
44 adults (aged between 18 and 65) with acute (< 6 weeks) unilateral symptomatic RC tendinopathy will be recruited.This single-blind (assessor), parallel-group RCT will include three evaluation sessions over 6 weeks (baseline, week 2, week 6) and one meeting with the treating physiotherapist (right after the baseline evaluation). All participants will take part in the baseline evaluation. They will first complete a questionnaire on sociodemographic, symptomatology and comorbidity, as well as self-administered questionnaires that evaluate symptoms and functional limitations (DASH, WORC and BPI). Then, ultrasonographic (US) measurements of AHD and of the supraspinatus tendon and subacromial bursal thickness will be conducted. Thereafter, pain inhibitory control will be assessed using conditioned pain modulation. Finally, the corticospinal excitability of the infraspinatus muscle will be evaluated. Thereafter, participants will be randomly assigned to one of two intervention groups, and then take part in their assigned home program. At week 2 and 6, the self-administered questionnaires will be re-administered (by phone for the week 6 evaluation). A global rating of change question (with % of change since baseline) will also be completed at week 2 and 6. US measurements, conditioned pain modulation and corticospinal excitability will only be revaluated at week 2. To evaluate the effectiveness of blinding, the assessor will complete a question related to his/her opinion of the allocation at week 2. The study will be carried out at the Centre interdisciplinaire de recherche en réadaptation et en intégration sociale (CIRRIS) by two different physiotherapists and in two different laboratories. Ethics approval will be obtained from Institutional Review Board of IRDPQ.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years old
* Acute (< 6 weeks) unilateral symptomatic rotator cuff tendinopathy
* Positive sign in each of the following categories: a) painful arc of movement, b) positive Neer or Kennedy-Hawkins tests, and c) pain on resisted isometric lateral rotation or abduction, or positive Jobe test.

Exclusion Criteria:

* Fracture at the symptomatic upper limb;
* Previous neck or shoulder surgery;
* Shoulder pain reproduced during active neck movement;
* Shoulder capsulitis;
* Clinical signs of a full thickness rotator cuff tear;
* Rheumatoid, inflammatory, or neurological diseases;
* Behavioural or cognitive problems.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand questionnaire | Change from baseline at 2 weeks, change from baseline at 6 weeks
  Generic questionnaire assessing any upper limb disorders

SECONDARY OUTCOMES:
Western Ontario Rotator Cuff index | Change from baseline at 2 weeks, change from baseline at 6 weeks
  Questionnaire specific to rotator cuff disorders
Short form of Brief Pain Inventory (questions 1-6 only) | Change from baseline at 2 weeks, change from baseline at 6 weeks
  Pain questionnaire
Acromiohumeral distance in cm using LogiqE9 (GE Healthcare, Milwaukee, WI, USA) ultrasound scanner | Change from baseline at 2 weeks
Supraspinatus tendon thickness in mm using LogiqE9 (GE Healthcare, Milwaukee, WI, USA) ultrasound scanner | Change from baseline at 2 weeks
Percentage change in pain perception using Conditioned Pain Modulation equipment | Change from baseline at 2 weeks
  This measurement represents the effectiveness of descending inhibitory mechanisms
Isometric shoulder external rotation strength | Change from baseline at 2 weeks
  Measured using hand-held digital dynamometer
Isometric shoulder abduction strength | Change from baseline at 2 weeks
  Measured using hand-held digital dynamometer
Shoulder flexion, external rotation at 0 degrees and 90 degrees abduction, internal rotation at 90 degrees abduction | Change from baseline at 2 weeks
  Measured using a digital inclinometer

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Interdisciplinary Research in Rehabilitation and Social Integration (CIRRIS), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dupuis F, Barrett E, Dube MO, McCreesh KM, Lewis JS, Roy JS. Cryotherapy or gradual reloading exercises in acute presentations of rotator cuff tendinopathy: a randomised controlled trial. BMJ Open Sport Exerc Med. 2018 Dec 26;4(1):e000477. doi: 10.1136/bmjsem-2018-000477. eCollection 2018. PMID 30622733